CLINICAL TRIAL: NCT01425047
Title: Bioavailability and Anti-inflammatory Activities of Mangostins: a Pilot Study
Brief Title: Bioavailability of Xanthones From Mangosteen
Status: Completed | Type: Observational
Sponsor: Mark Failla (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor-Investigator, Mark Failla, Professor, Human Nutrition, Associate Dean for Research, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2010H0219
Record Dates: First submitted 2011-08-26; First posted 2011-08-29 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Healthy Volunteers
Keywords: mangosteen; xanthones; dietary supplement; botanical supplement; bioavailability; Determine bioavailability of mangosteen xanthones in adults

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sera and urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Females ingesting mangosteen juice
- Males ingesting mangosteen juice

SUMMARY:
Mangosteen is a tropical tree. The peel of mangosteen fruit is used in traditional medicine. The purpose of this study was to determine the bioavailability of the xanthones from mangosteen juice in adult human subjects.

DETAILED DESCRIPTION:
Garcinia mangostana L. (mangosteen) is a tropical tree native to Southeast Asia. The pericarp of mangosteen fruit is used in traditional medicine to treat inflammation, infections, wounds, and diarrhea. The proposed health-promoting effects have been attributed to a family of polyphenols referred to as xanthones. Since its introduction into the United States, juices and products containing mangosteen fruit have become a top-selling botanical dietary supplement. This commercial success largely has been the result of aggressive marketing of health claims based on in vitro observations and anecdotal reports.

The purpose of this study was to determine the bioavailability of xanthones from mangosteen juice in adult human subjects. After an overnight fast of at least 10h, male and female subjects were admitted to the Ohio State University Clinical Research Center. Volunteers ingested 2 ounces of 100% mangosteen juice as part of a western-style breakfast. Pericarp particles accounted for 1% of the mass and 99% of total xanthone content in the juice. This dose provided 130 ± 2 mg total xanthones. Blood was collected prior to breakfast and 1,2,3,4,6,8 and 24h. Subjects were fed a mangosteen-free lunch and released from the unit after the 8h collection, refraining from mangosteen containing products until final collection of blood at 24h. Urine was collected for the 24 test period.

ELIGIBILITY:
Inclusion Criteria:

* 5 female
* 5 male
* body mass index </= 30
* normal renal function
* non-smoking

Exclusion Criteria:

* smokers
* acute or chronic diseases
* history of gastrointestinal diseases
* >/= 10% weight loss
* dietary or herbal supplement within 6 months of study
* pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 5 female and 5 male healthy, non-smoking subjects admitted to the Clinical Research Center at The Ohio State University.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-11; Primary Completion 2010-11 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Xanthones in urine | 0-24 hours
  Urine was collected prior to ingesting mangosteen juice with breakfast and then from consumpotion of juice until 24h.

SECONDARY OUTCOMES:
Xanthones in sera | 0-24 hours
  Blood was collected prior to breakfast, and 1, 2, 3, 4, 6, 8 and 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mark Failla, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Clinical Research Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Chitchumroonchokchai C, Riedl KM, Suksumrarn S, Clinton SK, Kinghorn AD, Failla ML. Xanthones in mangosteen juice are absorbed and partially conjugated by healthy adults. J Nutr. 2012 Apr;142(4):675-80. doi: 10.3945/jn.111.156992. Epub 2012 Mar 7. PMID 22399525